CLINICAL TRIAL: NCT00276731
Title: Randomized Study of Radiotherapy in Patients With Stage 2B/3 (INSS) Neuroblastoma in Children Over 1 Year of Age
Brief Title: Combination Chemotherapy Followed By Surgery With or Without Radiation Therapy in Treating Young Patients With Stage II or Stage III Neuroblastoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000454725; CCLG-NB-1995-02; EU-20595; UKCCSG-ENSG-9
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-01

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; localized unresectable neuroblastoma; regional neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cisplatin; Cyclophosphamide; Etoposide; Vincristine; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: vincristine sulfate
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain. It is not yet know whether combination chemotherapy followed by surgery alone is more effective than combination chemotherapy followed by surgery and radiation therapy in treating neuroblastoma.

PURPOSE: This randomized phase III trial is studying combination chemotherapy followed by surgery to see how well it works compared to combination chemotherapy followed by surgery and radiation therapy in treating young patients with stage II or stage III neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the local control and event-free and overall survival of young patients with stage IIB and III neuroblastoma treated with neoadjuvant combination chemotherapy followed by surgery with vs without radiotherapy.
* Determine the toxic effects of these regimen in these patients.

OUTLINE: This is a multicenter, randomized study.

* Induction combination chemotherapy: Patients receive vincristine IV and cyclophosphamide IV on day 1. Patients also receive cisplatin IV continuously over 24 hours on day 1 and etoposide IV over 4 hours on day 2 during courses 1, 3, and 5 and carboplatin IV over 1 hour and etoposide IV over 4 hours on day 1 during courses 2 and 4. Treatment repeats every 21 days for 5 courses in the absence of disease progression or unacceptable toxicity. Patients then proceed to surgery unless complete resection was done during initial staging and complete response was maintained.
* Surgery: Patients undergo biopsy or surgical resection of the tumor 2-3 weeks after completion of induction combination chemotherapy.
* Post-surgical treatment: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive two additional courses of combination chemotherapy comprising vincristine, cisplatin, etoposide, and cyclophosphamide in course 6 and vincristine, carboplatin, etoposide, and cyclophosphamide in course 7.
  * Arm II: Patients undergo radiotherapy 2-4 weeks after surgery. Beginning 3 weeks after completion of radiotherapy, patients receive chemotherapy as in arm I After completion of study treatment, patients are evaluated periodically.

PROJECTED ACCRUAL: A total of 150 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IIB or III neuroblastoma

  * No n-myc amplification

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-03

CONTACTS AND LOCATIONS:
Overall Officials: Ann Barrett, Study Chair — University of Glasgow; S. J. Keith Holmes, DO — St. George's Hospital; Janice A. Kohler, MD, FRCP — University Hospital Southampton NHS Foundation Trust; Andrew David J. Pearson, MD, FRCP, DCh — University of Newcastle Upon-Tyne; Jack van Hoff, MD — Yale University; Robert P. Castleberry, MD — University of Alabama at Birmingham; Kevin Murray, MD — Mercy Regional Cancer Center at Mercy Medical Center
Locations (22):
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales